CLINICAL TRIAL: NCT04665388
Title: LANDscape MApping of Epitopes and T Cell Receptors for Selected Cancers
Acronym: LANDMARC
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: LANDMARC
Record Dates: First submitted 2020-12-03; First posted 2020-12-11 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
Keywords: Epstein-Barr Virus related cancer; Human Papilloma Virus related cancer; Hepatocellular Carcinoma; solid tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- EBV-related cancer cohort: up to N=30
- HPV-related cancer cohort: up to N=45
- HCC cohort: up to N=30

SUMMARY:
This is a correlative research project aimed at characterizing the T cell mediated immune responses to hepatocellular carcinoma (HCC), as well as Epstein-Barr virus (EBV)- and human papillomavirus (HPV)-related cancers. This study will enroll approximately 105 patients over 48 months. Of these 105 patients, 30 are EBV-related cancer, 45 are HPV-related cancer, and 30 are HCC. Patients will have blood samples collected one time to identify cancer specific T cells and T cell receptors in their blood. They will also have tissue samples collected one time to study the different types of immune cells, especially the T cells and their receptors.

The 105 patients enrolled in this study will be compared to retrospective samples (N=210; 30 from EBV-related cancer cohort, 180 from HPV-related cancer cohort).

DETAILED DESCRIPTION:
The cloning of genes encoding the T cell receptor (TCR), the identification of tumor-associated antigens and the subsequent characterization of the first HLA-restricted T cell-defined antigenic epitope, were key findings illustrating direct recognition of cancer cells by T cells. These discoveries provided a mechanistic foundation for ensuing work examining the dynamic nature of lymphocyte-dependent recognition and elimination of neoplastic cells. Furthermore, preclinical and clinical investigations illustrate an important role for T cell mediated anti-tumor immunity in human disease, and have characterized the complexity of cancer-associated immune responses that are not always sufficient for tumor elimination. Importantly however, therapeutic targeting of the immune system has demonstrated the power of immunomodulatory drugs for the restoration of anti-tumor immune responses for cancer treatment.

Presence of lymphocytes in a variety of human cancers is well documented, and T cells isolated from tumors that recognize cancer antigens can be harnessed for effective treatment. T cells isolated from patient tumors can be ex vivo expanded, and reinfused back into patients in a regime of cellular therapy termed adoptive cell transfer (ACT). This ACT therapy can be further directed to specific tumor antigens with the genetic manipulation of T cells to express TCR recognizing known p-HLA epitopes with dominant expression on cancer cells. However, the peptide-HLA (p-HLA) epitope landscape of tumor associated antigens, and their cognate TCR are not well described, and those which have been described are primarily limited to the class I HLA-A*02:01 allele dominant only in European-Caucasian populations. The purpose of this study is to further document the cancer epitope landscape and provide a comprehensive characterization of TCR specificities in a range of malignancies, for a wide variety of class I and class II HLA alleles. In addition, we aim to elucidate not only TCR repertoires important for anti-tumor immunity, but further clarify the role antigen presenting cells play in shaping these T cell repertoires.

The objectives involve the identification of cancer-associated/specific antigen p-HLA epitopes and their cognate TCR, and the subsequent structural and functional characterization these TCR. To meet this objective, immune cells of T, B and myeloid lineage will be analyzed. Phenotypic characterization of these cell subsets will be performed using standard immunological procedures such as immunofluorescence, immunohistochemistry, ELISA, ELISpot, qRT-PCR, analytic cytometry, CyTOF (cytometry time of flight), and in vitro stimulation. To relate immune responses to cancer cell intrinsic biology, RNA and DNA will be sequenced to identify cancer cell transcriptome and mutations, as well as T cell receptor unique sequences. Results from all laboratory analysis will be combined with relevant clinical data. Any confirmation of diagnosis, tissue types and other clinical data will be provided as available from the pathologists of the relevant disease site at UHN.

An incomplete understanding of T cell responses to cancer impedes the development of more effective immunotherapeutics. Discovery using tumor specimens from cancer patients will clarify how the complexity of the tumor environment shapes T cell specificity to induce effective immune responses and facilitate our development of better immune modulating therapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histological or cytological diagnosis of:

   1. EBV-related malignancies (e.g. nasopharyngeal cancer)
   2. HPV-related malignancies, including squamous cell carcinoma of the head and neck, cervix, vulva or anal canal. HPV positivity is required for squamous cell cancers of the head and neck.; p16 positivity as a surrogate for HPV testing is acceptable. HPV positivity is not required for cervix, vulva or anal canal cancer.

      * For cancers of the anal canal, late stage distant metastatic tumor tissue is preferred. However, early stage primary site tissue is acceptable, if the tissue can be procured without contamination by intestinal microbiota.
   3. For HCC, only patients who have above UHN institutional upper limit of normal levels of alpha-fetoprotein (AFP) in serum will be eligible. The diagnosis of HCC should be made based on standard of care with or without tumor tissue confirmation.
2. Patients must be ≥ 18 years old.
3. Patients must have provided voluntary written informed consent.

Exclusion Criteria:

1. Any condition that, in the opinion of the Investigator, would interfere with patient safety, or evaluation of the collected specimens and interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid tumor patients, including patients with hepatocellular carcinoma (HCC) patients and Epstein-Barr virus (EBV)- human papillomaviruses (HPV)-related cancers.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Identifying the p-HLA epitopes across diverse HLA alleles | 63 months
  To identify the p-HLA epitopes, we will examine a variety of clinically relevant tumor antigens, including alpha feto-protein (AFP) and carcinoembryonic antigen (CEA) in HCC, and canonical and cryptic protein antigens specific to the EBV-sequence and HPV-sequence open reading frames (ORFs).

SECONDARY OUTCOMES:
Characterizing tumor-antigen specific TCR repertoire diversity across diverse HLA alleles, and further provide a comprehensive functional analysis that identifies immunodominant epitopes important for tumor control | 63 months
  To characterize, we will map the landscape of anti-tumor TCR repertoire diversity, and characterize the functional heterogeneity of clonotypic T cell responses for the cancer-type specific antigens. Where tumor tissue is available, comprehensive comparative analysis of immune populations in the peripheral blood will accompany those analyses of tumor tissue. Peripheral blood samples will be used for the three specific endpoints, including; 1) assessment of the functionality, composition, relative percentage, and absolute number of various immune cell populations, 2) quantitation of soluble factors influencing immune cell function, and 3) a comprehensive phenotypic and functional characterization of tumor specific T cells in the periphery.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Han, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There may be data sharing in the future for potential collaborations with external researchers within the scope of the study objectives.